CLINICAL TRIAL: NCT06769698
Title: Phase II Randomized Study of Fianlimab Plus Cemiplimab Versus Cemiplimab Plus Placebo in First-Line Treatment of Participants With Recurrent or Metastatic (R/M) Head and Neck Squamous Cell Carcinoma (HNSCC) That Is Positive for PD-L1 Expression
Brief Title: A Study to See if Giving Fianlimab and Cemiplimab Together is Better Than Cemiplimab Alone at Treating Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3767-ONC-2431; 2024-517620-19-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Recurrent or Metastatic (R/M); Positive for Programmed Death Ligand 1 (PD-L1) Expression; Human Papillomavirus (HPV)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis | interventions — cemiplimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Approximately 60 participants with HPV (human papillomavirus) positive HNSCC. Randomized 1:1 to Fianlimab + Cemiplmab Fixed Dose Combination (FDC) versus Cemiplimab + Placebo.
  Interventions: Drug: FDC fianlimab+cemiplimab; Drug: Cemiplimab; Drug: Placebo
- Cohort 2 (Experimental): Approximately 60 participants with HPV negative HNSCC. Randomization is the same as in Cohort 1.
  Interventions: Drug: FDC fianlimab+cemiplimab; Drug: Cemiplimab; Drug: Placebo

INTERVENTIONS:
Drug: FDC fianlimab+cemiplimab — Fixed-Dose Combination (FDC) Administered per the protocol
  Other Names: REGN3767; REGN2810; Libtayo
Drug: Cemiplimab — Administered per the protocol
  Other Names: R2810; Libtayo
Drug: Placebo — Administered per the protocol

SUMMARY:
This study is researching an experimental drug called fianlimab (also called REGN3767), combined with a medication called cemiplimab compared against cemiplimab combined with placebo (a placebo looks like a treatment but does not contain any real medicine), collectively called "study drugs" in this form.

The study is focused on participants with head and neck cancers who have not been previously treated for head and neck cancer that has come back or spread to other parts of the body, referred to as recurrent or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC).

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* How much of each study drug is in the blood at different times
* Whether the body makes antibodies against the study drug(s) individually (which could make the study drugs less effective or could lead to side effects)
* Compatible research to better understand the study drugs and HNSCC

ELIGIBILITY:
Key Inclusion Criteria:

1. Have histologically confirmed (by local pathology) R/M HNSCC that is considered incurable by local therapies
2. Primary tumor location of oral cavity, oropharynx, larynx, or hypopharynx (patients with cervical neck node SCC with occult primary as described in the protocol
3. PD-L1 expression Combined Positive Score (CPS) ≥1 documented with a previously PD-L1 obtained Immunohistochemistry (IHC) result prior to screening, as described in protocol
4. Oropharynx cancer participants only: HPV status, based on a previously documented result prior to screening, must have been established in a surgical biopsy specimen or a core biopsy specimen as described in the protocol
5. At least 1 lesion that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as described in the protocol
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Adequate organ and bone marrow function as described in the protocol

Key Exclusion Criteria:

Medical Conditions

1. Participants who have Progressive Disease (PD) within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC as described in the protocol
2. Participants who have a primary tumor site of nasopharynx, paranasal sinus or salivary gland (any histology)
3. Head and neck SCC with unknown primary site as described in the protocol
4. Participants with active, known, or suspected autoimmune disease that has required systemic therapy within 5 years of the projected enrollment date as described in the protocol
5. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management
6. History or current evidence of significant cardiovascular disease including, myocarditis, congestive heart failure (as defined by New York Heart Association Functional Classification III and IV), unstable angina, serious uncontrolled arrhythmia, and myocardial infarction 6 months prior to study enrollment.

   Prior/Concomitant Therapy
7. Participants who have received prior systemic anticancer therapy in the R/M HNSCC setting as described in the protocol
8. Participants with a condition requiring corticosteroid therapy (>10 mg prednisone/prednisolone/day or equivalent) within 14 days of the first dose of study drug as described in the protocol

Note: Other protocol defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-06-04 (Estimated); Study Completion 2030-12-28 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 90 days after last study treatment, approximately 58 months

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 90 days after last study treatment, approximately 58 months
Severity of AEs | Up to 90 days after last study treatment, approximately 58 months
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to 90 days after last study treatment, approximately 58 months
Incidence of immune-mediated Adverse Events (imAEs) | Up to 90 days after last study treatment, approximately 58 months
Incidence of treatment-related AEs | Up to 90 days after last study treatment, approximately 58 months
Incidence of Adverse Events of Special Interest (AESIs) | Up to 90 days after last study treatment, approximately 58 months
Incidence of Serious Adverse Events (SAEs) | Up to 90 days after last study treatment, approximately 58 months
Incidence of AEs leading to discontinuation | Up to 90 days after last study treatment, approximately 58 months
Incidence of AEs leading to death | Up to 90 days after last study treatment, approximately 58 months
Incidence of laboratory abnormalities | Up to 90 days after last study treatment, approximately 58 months
  Per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Disease Control Rate (DCR) per investigator assessment | Up to 90 days after last study treatment, approximately 58 months
Duration of Response (DOR) per investigator assessment or death, whichever occurs first | Up to 90 days after last study treatment, approximately 58 months
Progression-Free Survival (PFS) per investigator assessment or death, whichever occurs first | Up to 90 days after last study treatment, approximately 58 months
Concentrations of cemiplimab in serum | Up to 90 days after last study treatment, approximately 58 months
Concentrations of fianlimab in serum | Up to 90 days after last study treatment, approximately 58 months
Incidence of Anti-Drug Antibody (ADA) to fianlimab | Up to 90 days after last study treatment, approximately 58 months
Titer of ADA to fianlimab | Up to 90 days after last study treatment, approximately 58 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/